CLINICAL TRIAL: NCT03639753
Title: Promoting Transportation Safety in Adolescence
Brief Title: Transportation Safety in Adolescence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Edinburgh (Other); University of Alabama at Birmingham (Other); Children's Hospital of Philadelphia (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Catherine McDonald, PI, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-834765; R01HD095248 (NIH)
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Automobile Accident
Keywords: teen driver safety; injury prevention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-Teen Intervention (Experimental): Parent health coaching session and supportive materials, teen on road driver assessment with feedback.
  Interventions: Behavioral: Parent-Teen Intervention
- Usual Practice (Other)
  Interventions: Other: Usual Practice

INTERVENTIONS:
Behavioral: Parent-Teen Intervention — Parent health coaching and resources + teen on-road driver experience + safe driving eLearning Modules
  Arms: Parent-Teen Intervention
Other: Usual Practice — Standard care for teens who get licensed in the state of PA
  Arms: Usual Practice

SUMMARY:
The proposed project will focus on improving teen driver safety as motor vehicle crashes are the leading cause of death and injury to adolescents. If successful, research findings will lead to clear strategies to reduce motor vehicle crashes.

ELIGIBILITY:
Inclusion Criteria:

* Teens between 16 and 17 years and 4 months (17.33 years) of age
* Pennsylvania state learner's permits
* Will have their Pennsylvania state learner's permit for at least 6 months (self-report)
* Self-report of less than 10 hours of behind-the-wheel driving experience.
* Teen and parent/caregiver fluent in written and spoken English
* Access to at least one practice vehicle
* Email address and internet access to complete study procedures

Exclusion Criteria:

* Teens with self-reported or parent reported (of teen's) visual, medical, or physical impairments that would require a handicap placard or assistive device to drive.
* Teens with pervasive developmental delays
* Have a sibling enrolled in this study
* Enrolled in other teen driving studies

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2216 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Police-reported motor vehicle crashes | Baseline to 12 months after licensure
  Time to first motor vehicle crash

CONTACTS AND LOCATIONS:
Overall Officials: Leann Long, PhD, Principal Investigator — Wake Forest University Health Sciences; Catherine McDonald, PhD, RN, FAAN, Principal Investigator — University of Pennsylvania; Jessica Mirman, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Hafetz J, McDonald CC, Long DL, Ford CA, Mdluli T, Weiss A, Felkins J, Wilson N, MacDonald B. Promoting transportation safety in adolescence: the drivingly randomized controlled trial. BMC Public Health. 2023 Oct 17;23(1):2020. doi: 10.1186/s12889-023-16801-6. PMID 37848929